CLINICAL TRIAL: NCT01985542
Title: The Molecular Biological Effects of Immunotherapy in the Nose
Brief Title: The Effects of Immunotherapy in the Nose
Acronym: Birch11
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other); Finnish Institute of Occupational Health (Other)
Responsible Party: Principal Investigator, Sanna Salmi, MD PhD, Docent, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: The effects of immunotherapy
Record Dates: First submitted 2013-11-04; First posted 2013-11-15 (Estimated); Results first posted 2021-04-20 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Rhinitis, Allergic, Seasonal
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- subcutaneous immunotherapy (Active Comparator): Starts with birch pollen subcutaneous immunotherapy
  Interventions: Drug: birch pollen subcutaneous immunotherapy
- no immunotherapy (No Intervention): not starting with birch pollen subcutaneous immunotherapy

INTERVENTIONS:
Drug: birch pollen subcutaneous immunotherapy — birch pollen subcutaneous immunotherapy
  Arms: subcutaneous immunotherapy

SUMMARY:
Allergic rhinitis might be caused by decreased resistance of nasal barrier to allergens and other environmental insults. About 20 % of the European population suffers from pollen allergies. Birch pollen allergic rhinitis is the most common allergic disease in the Scandinavia and it exists widely also in the Central Europe. Suffering and high costs of pollen allergies may be reduced by understanding the molecular biology of the nasal barriers during allergic response. Our aim is to observe the effect of season and birch pollen immunotherapy on the molecular biology of nasal epithelium and the microbiome.

DETAILED DESCRIPTION:
This is a controlled study with an intervention arm, and a control group of healthy volunteers. The population is composed of nonsmoking healthy adults and patients having birch or timothy pollen allergy with rhinoconjuctivitis symptoms and without other diseases. The diagnosis of pollen allergy is verified with positive history, skin prick test, and allergen specific IgE antibodies. Subjects undergo a spirometry with a bronchodilatator test and a histamine challenge. Quality of life and patient history data is collected by questionnaires. Four peripheral blood samples, as well as nasal cell swabs from nasal mucosa without local anesthesia are collected from each patient; in spring and winter before the group of the intervention arm starts with birch pollen subcutaneous immunotherapy; and during the first spring and winter when a subgroups has received the birch pollen immunotherapy. We plan to perform the following analyses for the nasal specimens: transcriptomics and their regulators, sequencing of 16SrRNA and RT-qPCR for assessing mucosal microbiome, mass spectrometry for analyses of proteins and protein-protein complexes, immunohistochemistry for tissue level localization and quantitation of proteins, in silico analyses for the data mining, integration and display. In addition we observe the alterations in inflammatory mediators after in vitro allergen activation of purified peripheral blood leukocytes by ELISA and real time qPCR.

ELIGIBILITY:
Inclusion Criteria:

* allergic rhinoconjunctivitis of birch pollen OR healthy controls

Exclusion Criteria:

* smoking, asthma, any other disease than allergic rhinoconjunctivitis, requiring constant medication

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2011-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanna K Salmi, MD PhD, Principal Investigator — Helsinki University Central Hospital

IPD SHARING:
Plan to Share IPD: No
The individual participant data is not shared.

REFERENCES:
- [Background] Mattila P, Renkonen J, Toppila-Salmi S, Parviainen V, Joenvaara S, Alff-Tuomala S, Nicorici D, Renkonen R. Time-series nasal epithelial transcriptomics during natural pollen exposure in healthy subjects and allergic patients. Allergy. 2010 Feb;65(2):175-83. doi: 10.1111/j.1398-9995.2009.02181.x. Epub 2009 Oct 5. PMID 19804444
- [Background] Joenvaara S, Mattila P, Renkonen J, Makitie A, Toppila-Salmi S, Lehtonen M, Salmi P, Lehti S, Makinen J, Sormunen R, Paavonen T, Renkonen R. Caveolar transport through nasal epithelium of birch pollen allergen Bet v 1 in allergic patients. J Allergy Clin Immunol. 2009 Jul;124(1):135-142.e1-21. doi: 10.1016/j.jaci.2008.11.048. Epub 2009 Apr 2. PMID 19344938

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subcutaneous Immunotherapy | no Immunotherapy
Started | 7 | 9
Completed | 3 | 3
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Population: Immunotherapy group is starting with subcutaneuous birch pollen immunotherapy (AIT) with normal protocol of the Hospital. Control group is not starting AIT.
Groups:
- Subcutaneous Immunotherapy: Starting with subcutaneuous birch pollen immunotherapy with normal protocol of the Hospital
- no Immunotherapy: Birch pollen allergic subjects that are not starting with immunotherapy
- Total: Total of all reporting groups
Arm/Group | Subcutaneous Immunotherapy | no Immunotherapy | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants] — Volunteers
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 3 | 3 | 6
    >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 40 [37 to 45] | 34 [30 to 49] | 38.5 [30 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  Finland | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: The Total Number of Differentially Expressed Transcripts.
Description: Transcriptomics are evaluated By Next Generation Sequencing. The total number of differentially expressed transcripts are defined from nasal epithelial brushing samples taken at -6 months vs. at +6 months in the two subject groups.
  The subject groups are the Subcutaneous immunotherapy group and No immunotherapy group.
Time Frame: -6 months vs. +6 months from the starting point of birch pollen subcutaneous immunotherapy.
Measure: Number; unit: transcripts
Units Other Than Participants: nasal brushing sample
Groups:
- Subcutaneous Immunotherapy; No Immunotherapy: Subjects with birch pollen allergic rhinitis.
Arm/Group | Subcutaneous Immunotherapy | No Immunotherapy
Number analyzed (Participants) | 3 | 3
Number analyzed (nasal brushing sample) | 6 | 6
transcripts | 119 | 49

2. Secondary Outcome: Percentage Change in Visual Analogue Scale Scores of Symptoms
Description: Visual analogue scale (VAS) was measured as 0-100 mm per each symptom question. VAS value 0 (mm) indicates no symptoms, and value 100 (mm) indicates the worst case.
  Total VAS score = sum of the VAS scores for the 41 symptoms The minimum value of the total VAS score is 0, and the maximum value is 4100. Relative change = [(measure at time +6 months - measure at time -6 months)]/measure at time -6 months * 100%.
  Measure = total VAS score
Time Frame: -6 months vs. +6 months from the starting point of birch pollen subcutaneous immunotherapy.
Population: The subject groups are the Subcutaneous immunotherapy group and No immunotherapy group.
Measure: Median (Full Range); unit: percent change
Groups:
- Immunotherapy; No Immunotherapy: Subjects with birch pollen allergic rhinitis.
Arm/Group | Immunotherapy | No Immunotherapy
Number analyzed (Participants) | 3 | 3
percent change | -68 [-76 to -7] | 91 [-49 to 347]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 18 months
Description: Interview and marking to Immunotherapy form of the patient records.
Arm/Group | Subcutaneous Immunotherapy | no Immunotherapy
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/9
Other Adverse Events (participants affected / at risk) | 0/7 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No